CLINICAL TRIAL: NCT04613596
Title: A Phase 2 Trial of Adagrasib Monotherapy and in Combination With Pembrolizumab and a Phase 3 Trial of Adagrasib in Combination With Pembrolizumab Versus Pembrolizumab in Patients With Advanced Non-Small Cell Lung Cancer With KRAS G12C Mutation
Brief Title: Phase 2 Trial of Adagrasib Monotherapy and in Combination With Pembrolizumab and a Phase 3 Trial of Adagrasib in Combination in Patients With a KRAS G12C Mutation KRYSTAL-7
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0009; CA239-0009 (Other: Bristol-Myers Squibb Protocol ID); 849-007 (Other: Mirati Therapeutics Protocol ID)
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Advanced Non-Small Cell Lung Cancer; Metastatic Non-Small Cell Lung Cancer
Keywords: KRAS G12C; Non-small cell lung cancer; NSCLC; Metastatic Non-Small Cell Lung Cancer; Adagrasib; Krazati; TPS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — adagrasib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: MRTX849 Monotherapy, MRTX849 in Combination with Pembrolizumab and Pembrolizumab alone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 2 Cohort 1a: PD-L1 TPS <1% (Experimental): Cohort 1a: Adagrasib twice daily (BID) in combination with pembrolizumab
  Interventions: Drug: Adagrasib
- Phase 2 Cohort 1b: PD-L1 TPS <1% (Experimental): Cohort 1b: Adagrasib BID monotherapy
  Interventions: Drug: Adagrasib
- Phase 2 Cohort 2: PD-L1 TPS ≥1% (Experimental): Cohort 2: Adagrasib BID in combination with pembrolizumab
  Interventions: Drug: Adagrasib
- Phase 3 Cohort 3 Investigational Arm (Experimental): Adagrasib BID in combination with pembrolizumab
  Interventions: Drug: Adagrasib
- Phase 3 Cohort 4 Comparator Arm (Active Comparator): Pembrolizumab
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Adagrasib — Adagrasib 400 mg twice daily (BID) in combination with pembrolizumab (Cohort 1a)
  Other Names: Pembrolizumab
  Arms: Phase 2 Cohort 1a: PD-L1 TPS <1%
Drug: Adagrasib — Adagrasib 600 mg BID monotherapy (Cohort 1b)
  Arms: Phase 2 Cohort 1b: PD-L1 TPS <1%
Drug: Adagrasib — adagrasib 400 mg BID in combination with pembrolizumab
  Other Names: Pembrolizumab
  Arms: Phase 2 Cohort 2: PD-L1 TPS ≥1%
Drug: Adagrasib — Adagrasib 400 mg BID + pembrolizumab 200 mg every Q3W
  Other Names: Pemrolizumab
  Arms: Phase 3 Cohort 3 Investigational Arm
Drug: Pembrolizumab — Pembrolizumab 200 mg IV Q3W
  Arms: Phase 3 Cohort 4 Comparator Arm

SUMMARY:
The Phase 2 portion of this study evaluates the efficacy and safety of MRTX849 monotherapy and in combination with pembrolizumab in cohorts of patients with advanced NSCLC with KRAS G12C mutation and any PD-L1 TPS and who are candidates for first-line treatment.

The Phase 3 portion of the study compares the efficacy of adagrasib in combination with pembrolizumab versus pembrolizumab in patients with unresectable, locally advanced or metastatic squamous or nonsquamous NSCLC with KRAS G12C mutation and PD-L1 TPS >=50% and who are candidates for first line treatment.

DETAILED DESCRIPTION:
The Phase 2 portion of this study will evaluate the efficacy and safety of MRTX849 as monotherapy and in combination with pembrolizumab. There will be 3 cohorts of patients, all of whom have KRAS G12C mutation, have advanced or metastatic NSCLC, and are candidates for first-line treatment. 2 cohorts have PD-L1 TPS score <1% and are randomized to MRTX849 monotherapy or MRTX849 in combination with pembrolizumab. The 3rd cohort has PD-L1 TPS score of 1% or higher and is treated with MRTX849 and pembrolizumab

The Phase 3 portion of the study will randomize patients with squamous or nonsquamous NSCLC with KRAS G12C mutation and TPS >=50% in the first-line setting to adagrasib plus pembrolizumab or pembrolizumab. Primary efficacy objective is to compare efficacy between experimental and comparator arms. Secondary and exploratory objectives include evaluation of secondary efficacy endpoints, safety and tolerability, adagrasib PK, PROs, and correlative genomic biomarkers for the combination regimen in the study population.

MRTX849 is an orally available small molecule inhibitor of KRAS G12C, and Pembrolizumab (KEYTRUDA®) is a humanized monoclonal antibody that blocks the interaction between PD-1 and its ligands, PD-L1 and PD-L2.

ELIGIBILITY:
Inclusion Criteria:

* Phase 2: Histologically confirmed diagnosis of unresectable or metastatic NSCLC with KRAS G12C mutation and any PD-L1 TPS
* Phase 3: Histologically confirmed diagnosis of unresectable or metastatic squamous or nonsquamous NSCLC with KRAS G12C mutation and PD-L1 TPS >=50%
* Phase 3: Presence of evaluable or measurable disease per RECIST
* Phase 3: CNS Inclusion - Based on screening brain imaging, patients must have one of the following:

  1. No evidence of brain metastases
  2. Untreated brain metastases not needing immediate local therapy
  3. Previously treated brain metastases not needing immediate local therapy

Exclusion Criteria:

* Phase 2 and Phase 3: Prior systemic treatment for locally advanced or metastatic NSCLC including chemotherapy, immune checkpoint inhibitor therapy, or a therapy targeting KRAS G12C mutation (e.g., AMG 510).
* Phase 2: Active brain metastases
* Phase 3: Patients with known central nervous system (CNS) lesions must not have any of the following:

  1. Any untreated brain lesions > 1.0 cm in size
  2. Any brainstem lesions
  3. Ongoing use of systemic corticosteroids for control of symptoms of brain lesions at a total daily dose of > 10 mg of prednisone (or equivalent) prior to randomization.
  4. Have poorly controlled (> 1/week) generalized or complex partial seizures, or manifest neurologic progression due to brain lesions notwithstanding CNS-directed therapy
* Phase 3: Radiation to the lung > 30 Gy within 6 months prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Phase 2: To evaluate the efficacy of Adagrasib monotherapy and in combination with pembrolizumab administered to patients having advanced/metastatic NSCLC. | 22 months
  Objective Response Rate (ORR) as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
Phase 3: To compare efficacy of Adagrasib in combination with pembrolizumab versus pembrolizumab | 36 months
  Progression Free Survival per RECIST 1.1 by Blinded Independent Central Review (BICR) and Overall Survival

SECONDARY OUTCOMES:
Phase 2: To characterize the safety and tolerability of study treatments in selected populations | 22 months
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of adverse events and laboratory abnormalities.
Phase 2: Duration of Response | 22 months
  Defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of either Progression of Disease (PD) or death due to any cause, whichever occurs first.
Phase 2: Progression Free Survival | 22 months
  Defined as time from first study treatment until disease progression or death from any cause, whichever occurs first.
Phase 2: To evaluate secondary efficacy endpoints using the study treatment in selected populations | 12 months
  1-Year Survival rate
Phase 2: To evaluate secondary efficacy endpoints using the study treatment in selected populations | 22 months
  Overall Survival (OS)
Phase 2: To evaluate the pharmacokinetics (PK) of study treatments by measuring blood plasma MRTX849 and potential metabolite concentrations. | 22 months
  Pharmacokinetics (PK) Blood plasma Adagrasib and potential metabolite concentrations
Phase 3: To evaluate the safety and tolerability in the study population | 36 months
  Safety characterized by type, incidence, severity, timing, seriousness and relationship to study treatment of adverse events and laboratory abnormalities.
Phase 3: To evaluate the PK of adagrasib administered in the study population | 36 months
  Pharmacokinetics (PK) Blood plasma Adagrasib and potential metabolite concentrations
Phase 3: To evaluate health-related quality of life (HRQOL) and lung cancer specific symptoms in the study population | 36 months
  Patient Reported Outcomes to measure quality of life
Phase 3: Progression Free Survival per RECIST 1.1 by Investigator | 36 months
  Defined as time from first study treatment until disease progression or death from any cause, whichever occurs first.
Phase 3: Duration of Response (DOR) per RECIST 1.1 by Investigator and BICR | 36 months
  Defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of either Progression of Disease (PD) or death due to any cause, whichever occurs first.
Phase 3: Objective Response Rate (ORR) per RECIST 1.1 by Investigator and BICR | 36 months
  Defined as the percent of patients documented to have a confirmed CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (755):
- United States (220):
  - Local Institution - 007-556-A, Goodyear, Arizona
  - USOR - Arizona Oncology - Prescott Valley, Prescott Valley, Arizona
  - Local Institution - 007-568-A, Safford, Arizona
  - Local Institution - 007-568-B, Safford, Arizona
  - Local Institution - 007-568-C, Safford, Arizona
  - Local Institution - 007-568-D, Safford, Arizona
  - Local Institution - 007-568-E, Safford, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Highlands Oncology Group - Springdale, Springdale, Arkansas
  - Providence - Saint Joseph Home Health - Anaheim, Anaheim, California
  - The Oncology Institute of Hope and Innovation - Corporate Office, Cerritos, California
  - Local Institution - 007-777, Fountain Valley, California
  - Local Institution - 007-778, Laguna Hills, California
  - Local Institution - 007-898-B, Long Beach, California
  - MemorialCare - Long Beach Medical Center, Long Beach, California
  - TRIO - Cancer & Blood Specialty Clinic - Los Alamitos, Los Alamitos, California
  - Local Institution - 007-579, Los Angeles, California
  - Local Institution - Unk045, Rancho Mirage, California
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Local Institution - 007-898-C, Santa Ana, California
  - Providence Medical Group - Santa Rosa, Santa Rosa, California
  - Stockton Hematology Oncology Medical Group (SHOMG) - Stockton (Suite B), Stockton, California
  - Local Institution - 007-898-A, Whittier, California
  - Local Institution - 007-872-H, Aurora, Colorado
  - Local Institution - 007-872-D, Boulder, Colorado
  - Local Institution - 007-872-L, Centennial, Colorado
  - Local Institution - 007-872-C, Colorado Springs, Colorado
  - Local Institution - 007-872-K, Colorado Springs, Colorado
  - Local Institution - 007-872-E, Denver, Colorado
  - Local Institution - 007-872-I, Denver, Colorado
  - Local Institution - 007-872-A, Lakewood, Colorado
  - Local Institution - 007-872-J, Littleton, Colorado
  - USOR - Rocky Mountain Cancer Centers - Lone Tree, Lone Tree, Colorado
  - Local Institution - 007-872-G, Longmont, Colorado
  - Local Institution - 007-872-B, Pueblo, Colorado
  - Local Institution - 007-872-F, Thornton, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Local Institution - 007-5476, Washington D.C., District of Columbia
  - GenesisCare USA, Aventura, Florida
  - Bay Pines Veterans Affairs Healthcare System, Bay Pines, Florida
  - Local Institution - 007-922-A, Bonita Springs, Florida
  - Local Institution - 007-922-D, Bradenton, Florida
  - Local Institution - 007-922-E, Cape Coral, Florida
  - Local Institution - 007-896-A, Celebration, Florida
  - Local Institution - 007-926-B, Daytona Beach, Florida
  - Local Institution - 007-562-B, Fleming Island, Florida
  - SCRI - Florida Cancer Specialists - South Region Research Office, Fort Myers, Florida
  - Local Institution - 007-922-B, Fort Myers, Florida
  - Local Institution - 007-922-C, Fort Myers, Florida
  - 21st Century Oncology of Jacksonville - North Lee Street, Jacksonville, Florida
  - Local Institution - 007-562-D, Jacksonville, Florida
  - Local Institution - 007-562-E, Jacksonville, Florida
  - Local Institution - 007-562-G, Jacksonville, Florida
  - Local Institution - 007-829, Jacksonville, Florida
  - Cancer Specialists of North Florida - Southpoint, Jacksonville, Florida
  - Local Institution - 007-562-C, Jacksonville, Florida
  - Local Institution - 007-562-F, Jacksonville Beach, Florida
  - Miami Veterans Affairs Healthcare System, Miami, Florida
  - Local Institution - 007-922-F, Naples, Florida
  - Local Institution - 007-922-G, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - USOR - Woodlands Medical Specialists, Pensacola, Florida
  - Local Institution - 007-922-H, Port Charlotte, Florida
  - Local Institution - 007-562-A, Saint Augustine, Florida
  - Local Institution - 007-922-I, Sarasota, Florida
  - Local Institution - 007-922-J, Sarasota, Florida
  - Local Institution - 007-926-D, Stuart, Florida
  - Local Institution - 007-924-A, Tallahassee, Florida
  - SCRI - Florida Cancer Specialists - Tallahassee Cancer Center, Tallahassee, Florida
  - James A. Haley Veterans Hospital, Tampa, Florida
  - Local Institution - Unk065, Tampa, Florida
  - Local Institution - 007-922-L, Venice, Florida
  - Local Institution - 007-922-K, Venice, Florida
  - Local Institution - 007-926-C, Vero Beach, Florida
  - Local Institution - 007-926-A, Wellington, Florida
  - SCRI - Florida Cancer Specialists - West Palm Beach, West Palm Beach, Florida
  - Local Institution - Unk072, Weston, Florida
  - University Cancer & Blood Center (UCBC) - Athens, Athens, Georgia
  - Local Institution - Unk052, Atlanta, Georgia
  - Local Institution - 007-786-C, Carrollton, Georgia
  - Local Institution - 007-786-A, Cartersville, Georgia
  - Local Institution - 007-786-D, Douglasville, Georgia
  - Local Institution - 007-786-B, Hiram, Georgia
  - Central Georgia Cancer Care - Macon, Macon, Georgia
  - Northwest Georgia Oncology Centers Wellstar - Marietta, Marietta, Georgia
  - Local Institution - 007-897, Honolulu, Hawaii
  - Local Institution - Unk005, Honolulu, Hawaii
  - Local Institution - 007-883-A, Arlington Heights, Illinois
  - Local Institution - 007-955, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - USOR - Illinois Cancer Specialists - Niles, Niles, Illinois
  - Advocate Medical Group Oncology, Park Ridge, Illinois
  - Local Institution - Unk061, Peoria, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Local Institution - 007-942-B, Chanute, Kansas
  - Local Institution - 007-942-D, El Dorado, Kansas
  - Local Institution - 007-942-E, Independence, Kansas
  - Local Institution - 007-942-F, Kingman, Kansas
  - Local Institution - 007-942-G, Liberal, Kansas
  - Local Institution - 007-942-H, McPherson, Kansas
  - MidAmerica Cancer Care - Research, Merriam, Kansas
  - Local Institution - 007-942-I, Newton, Kansas
  - Local Institution - 007-942-J, Parsons, Kansas
  - Local Institution - 007-942-K, Pratt, Kansas
  - Local Institution - 007-942-L, Salina, Kansas
  - Local Institution - 007-942-M, Wellington, Kansas
  - Local Institution - Unk032, Westwood, Kansas
  - Local Institution - 007-942-A, Wichita, Kansas
  - Cancer Center of Kansas - Wichita - Heritage Plaza, Wichita, Kansas
  - Local Institution - 007-942-N, Winfield, Kansas
  - Lexington Medical Cancer Center Hematology/Oncology, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Local Institution - 007-388-A, Louisville, Kentucky
  - Local Institution - Unk011, Baton Rouge, Louisiana
  - Local Institution - 007-994-A, Covington, Louisiana
  - Pontchartrain Cancer Center - Covington Office, Covington, Louisiana
  - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute at St. Elizabeths Medical Center, Brighton, Massachusetts
  - Brigham and Womens/Mass General Health Care Center at Foxborough, Foxborough, Massachusetts
  - Dana-Farber Cancer Institute - Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber Brigham and Womens Cancer Center at Milford Regional, Milford, Massachusetts
  - Dana-Farber Brigham Cancer Center at South Shore Health, South Weymouth, Massachusetts
  - USOR - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Local Institution - 007-589A, Edina, Minnesota
  - Local Institution - Unk006, Minneapolis, Minnesota
  - Local Institution - 007-822, Minneapolis, Minnesota
  - Local Institution - 007-830, Rochester, Minnesota
  - Jackson Oncology Associates - The Hederman Cancer Center, Jackson, Mississippi
  - Local Institution - 007-590D, Grand Island, Nebraska
  - Local Institution - 007-590A, Omaha, Nebraska
  - Local Institution - 007-590B, Omaha, Nebraska
  - Nebraska Cancer Specialists - Midwest Cancer Center - Legacy, Omaha, Nebraska
  - Local Institution - 007-590C, Papillion, Nebraska
  - OptumCare Nevada, Las Vegas, Nevada
  - Local Institution - 007-938A, Las Vegas, Nevada
  - Local Institution - 007-938B, Las Vegas, Nevada
  - Local Institution - 007-993, Belleville, New Jersey
  - Astera Cancer Care - East Brunswick, East Brunswick, New Jersey
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Local Institution - 007-975-A, Somerset, New Jersey
  - Local Institution - 007-975-B, Somerset, New Jersey
  - Local Institution - 007-975-C, Somerset, New Jersey
  - Local Institution - 007-975-D, Somerset, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - New York Oncology Hematology - Albany Medical Center, Albany, New York
  - Local Institution - Unk077, Rhinebeck, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Local Institution - 007-893-B, Cincinnati, Ohio
  - USOR - Oncology Hematology Care - Blue Ash, Cincinnati, Ohio
  - Local Institution - 007-893-C, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Mark H. Zangmeister Cancer Center, Columbus, Ohio
  - Local Institution - 007-893-A, Fairfield, Ohio
  - Kettering Health Cancer Center - Main Campus, Kettering, Ohio
  - Tricounty Hematology and Oncology - Massillon, Massillon, Ohio
  - USOR - Willamette Valley Cancer Institute and Research Center - Eugene, Eugene, Oregon
  - Local Institution - 007-885B, Portland, Oregon
  - Local Institution - 007-885A, Portland, Oregon
  - Oregon Oncology Specialists, Salem, Oregon
  - Local Institution - 007-885C, Tigard, Oregon
  - Local Institution - Unk041, Allentown, Pennsylvania
  - Veterans Affairs Pittsburgh Healthcare System - University Drive Campus, Pittsburgh, Pennsylvania
  - Local Institution - 007-960, Providence, Rhode Island
  - Local Institution - Unk038, Charleston, South Carolina
  - Local Institution - 007-5475, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Local Institution - 007-928-L, Dickson, Tennessee
  - Local Institution - 007-928-J, Franklin, Tennessee
  - Local Institution - 007-928-G, Gallatin, Tennessee
  - West Cancer Center & Research Institute - East Campus, Germantown, Tennessee
  - Local Institution - 007-928-A, Hendersonville, Tennessee
  - Local Institution - 007-928-D, Hermitage, Tennessee
  - Local Institution - 007-928-H, Lebanon, Tennessee
  - Local Institution - 007-928-F, Murfreesboro, Tennessee
  - Local Institution - 007-928-B, Nashville, Tennessee
  - Tennessee Oncology - Nashville - Centennial Clinic - Medical Oncology, Nashville, Tennessee
  - Local Institution - 007-928-K, Nashville, Tennessee
  - Local Institution - 007-928-E, Nashville, Tennessee
  - Local Institution - 007-928-C, Nashville, Tennessee
  - Local Institution - 007-928-M, Shelbyville, Tennessee
  - Local Institution - 007-928-I, Smyrna, Tennessee
  - Local Institution - 007-554B, Abilene, Texas
  - Local Institution - 007-554G, Amarillo, Texas
  - Local Institution - 007-879-A, Arlington, Texas
  - Local Institution - 007-879-B, Arlington, Texas
  - Local Institution - 007-892-B, Austin, Texas
  - Local Institution - 007-892-A, Austin, Texas
  - USOR - Texas Oncology - Dallas Fort Worth (DFW) - South Austin, Austin, Texas
  - Local Institution - 007-879-C, Bedford, Texas
  - Local Institution - Unk059, Dallas, Texas
  - Local Institution - 007-592, Dallas, Texas
  - Texas Oncology - Dallas Fort Worth (DFW) - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - USOR - Texas Oncology Northeast Texas - Denison, Denison, Texas
  - Local Institution - 007-554E, El Paso, Texas
  - Local Institution - 007-554C, El Paso, Texas
  - Local Institution - 007-554F, El Paso, Texas
  - USOR - Texas Oncology - Fredericksburg, Fredericksburg, Texas
  - Local Institution - 007-848, Houston, Texas
  - Local Institution - 007-999, Irving, Texas
  - Local Institution - 007-890-B, Longview, Texas
  - Local Institution - 007-554A, Midland, Texas
  - USOR - Texas Oncology - Dallas Fort Worth (DFW) - Odessa West Texas Cancer Center, Odessa, Texas
  - USOR - Texas Oncology - The Woodlands, The Woodlands, Texas
  - Local Institution - 007-890-A, Tyler, Texas
  - Local Institution - 007-554D, Wichita Falls, Texas
  - Local Institution - 007-912, Salt Lake City, Utah
  - Local Institution - 007-814-A, Alexandria, Virginia
  - Local Institution - 007-814-D, Arlington, Virginia
  - USOR - Virginia Cancer Specialists - Fairfax Office, Fairfax, Virginia
  - Local Institution - 007-814-B, Gainesville, Virginia
  - Local Institution - 007-814-C, Leesburg, Virginia
  - Virginia Cancer Institute - West End, Richmond, Virginia
  - USOR - Northwest Cancer Specialists, P.C. dba Compass Oncology - Vancouver Cancer Center, Vancouver, Washington
  - Local Institution - Unk064, Huntington, West Virginia
  - Local Institution - Unk057, Madison, Wisconsin
  - Local Institution - Unk068, Madison, Wisconsin
- Argentina (11):
  - Local Institution - 007-5001, Belgrano, Buenos Aires
  - Fundacion Respirar, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - Unk043, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Argentino de Diagnostico y Tratamiento, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Centro Oncologico Korben, San Pedro, Buenos Aires
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Sanatorio Parque, Rosario, Santa Fe Province
  - Local Institution - Unk053, Buenos Aires
  - Instituto Oncologico de Cordoba (IONC), Córdoba
  - Local Institution - Unk033, Porto Alegre
  - Local Institution - Unk020, Río Cuarto
- Australia (8):
  - Ballarat Regional Integrated Cancer Center, Ballarat
  - Flinders Medical Centre, Bedford Park
  - Local Institution - 007-004, Clayton
  - Canberra Hospital, Garran
  - Icon Cancer Centre, Hyde Park
  - Port Macquarie Base Hospital, Port Macquarie
  - Cancer Care Wollongong, Wollongong
  - Princess Alexandra Hospital, Woolloongabba
- Austria (6):
  - Klinikum Klagenfurt Am Worthersee, Klagenfurt
  - Universitatsklinikum Krems, Krems
  - Ordensklinikum Linz Elisabethinen, Linz
  - Medizinische Universitat Wien, Vienna
  - Wiener Gesundheitsverbund - Klinik Hietzing, Vienna
  - Wiener Gesundheitsverbund - Klinik Floridsdorf, Vienna
- Belgium (4):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Local Institution - 007-152, Roeselare
- Brazil (10):
  - Local Institution - 007-458, Natal, Rio Grande do Norte
  - Local Institution - Unk050, Lajeado, Rio Grande do Sul
  - Local Institution - Unk015, Porto Alegre, Rio Grande do Sul
  - Local Institution - Unk060, Barretos
  - Local Institution - 007-457, Barretos
  - Local Institution - Unk002, Ijuí
  - Local Institution - 007-459, Porto Alegre
  - Local Institution - Unk003, Rio de Janeiro
  - Local Institution - Unk019, São José do Rio Preto
  - Local Institution - Unk074, São Paulo
- Bulgaria (5):
  - Multiprofile Hospital For Active Treatment - Dr. Tota Venkova, Gabrovo
  - Specialized Hospital for Active Oncology Treatment - Haskovo SLLC (SBALO - Haskovo - EOOD), Haskovo
  - Complex Oncology Center - Plovdiv - Base II, Plovdiv
  - University Multiprofile Hospital for Active Treatment St. Ivan Rilski, Sofia
  - Complex Oncology Center - Vratsa, Vratsa
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Vancouver, Vancouver, British Columbia
  - Local Institution - 007-489, London, Ontario
  - Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Local Institution - 007-490, Montreal, Quebec
- Chile (2):
  - Local Institution - Unk028, Santiago
  - Local Institution - Unk073, Temuco
- China (155):
  - Local Institution - 007-051, Bengbu, Anhui
  - The First Affiliated Hospital of Bengbu Medical College/Department of Respiratory and Critical Care Medicine, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Local Institution - 007-026-Ph2, Hefei, Anhui
  - Local Institution - 007-026, Hefei, Anhui
  - Local Institution - 007-739-Ph2, Hefei, Anhui
  - Local Institution - 007-739, Hefei, Anhui
  - Local Institution - 007-747, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences/Medical Oncology Department, Beijing, Beijing Municipality
  - Local Institution - 007-050, Beijing, Beijing Municipality
  - Local Institution - 007-707-Ph2, Beijing, Beijing Municipality
  - Local Institution - 007-707, Beijing, Beijing Municipality
  - Local Institution - 1025-Ph2, Beijing, Beijing Municipality
  - Local Institution - 1025, Beijing, Beijing Municipality
  - Beijing Cancer Hospital/Thoracic Oncology(2nd) Department, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Local Institution - 007-027-Ph2, Beijing, Beijing Municipality
  - Local Institution - 007-038-Ph2, Beijing, Beijing Municipality
  - Local Institution - 007-038, Beijing, Beijing Municipality
  - Local Institution - 007-040-Ph2, Beijing, Beijing Municipality
  - Local Institution - 007-040, Beijing, Beijing Municipality
  - Local Institution - 007-718-Ph3, Chongqing, Chongqing Municipality
  - Local Institution - 1029-Ph2, Chongqing, Chongqing Municipality
  - Local Institution - 1029, Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital/Respiratory Ward of Tumor Center, Chongqing, Chongqing Municipality
  - Local Institution - 007-053, Chongqing, Chongqing Municipality
  - Local Institution - 1046-Ph2, Fuzhou, Fujian
  - Local Institution - 1046, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Local Institution - 007-039-Ph2, Fuzhou, Fujian
  - Local Institution - 007-039, Fuzhou, Fujian
  - Local Institution - 007-714-Ph2, Xiamen, Fujian
  - Local Institution - 007-714, Xiamen, Fujian
  - Local Institution - 007-732-Ph2, Xiamen, Fujian
  - Local Institution - 007-732, Xiamen, Fujian
  - The First Affiliated Hospital of Xiamen University/Medical Oncology Department, Xiamen, Fujian
  - Local Institution - 1022-Ph2, Guangzhou, Guangdong
  - Local Institution - 1022, Guangzhou, Guangdong
  - Local Institution - 007-712-Ph2, Guangzhou, Guangdong
  - Local Institution - 007-712, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Local Institution - 007-705-Ph2, Guangzhou, Guangdong
  - Local Institution - 007-705, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University/Respiratory Medicine Department, Guangzhou, Guangdong
  - Local Institution - 007-052, Shenzhen, Guangdong
  - Shenzhen People's Hospital/Department of Respiratory and Critical Care Medicine, Shenzhen, Guangdong
  - Local Institution - 007-704-Ph2, Liuchow, Guangxi
  - Local Institution - 007-704, Liuchow, Guangxi
  - Guangxi Medical University Cancer Hospital/Department of Respiratory Oncology, Nanning, Guangxi
  - Local Institution - 007-384, Nanning, Guangxi
  - Local Institution - 007-744-Ph2, Nanning, Guangxi
  - Local Institution - 1038-Ph2, Nanning, Guangxi
  - Local Institution - 1038, Nanning, Guangxi
  - Local Institution - 007-742, Shijiazhuang, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Cancer Hospital affiliated to Harbin Medical University/Ward 3 of Respiratory Medicine Department, Harbin, Heilongjiang
  - Local Institution - 007-028-Ph2, Harbin, Heilongjiang
  - Local Institution - 007-028, Harbin, Heilongjiang
  - Local Institution - 1012-Ph2, Xinxiang, Henan
  - Henan Cancer Hospital/Second Ward of Respiratory Medicine Department, Zhengzhou, Henan
  - Local Institution - 007-730-Ph3, Zhengzhou, Henan
  - Local Institution - 1010-Ph2, Zhengzhou, Henan
  - Local Institution - 1010, Zhengzhou, Henan
  - Local Institution - 007-021-Ph2, Zhengzhou, Henan
  - Local Institution - 007-715-Ph2, Zhengzhou, Henan
  - Local Institution - 007-715, Zhengzhou, Henan
  - Local Institution - 007-730-Ph2, Zhengzhou, Henan
  - Local Institution - 007-719-Ph2, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology/Cancer Center Department, Wuhan, Hubei
  - Local Institution - 007-700-Ph2, Wuhan, Hubei
  - Local Institution - 007-700, Wuhan, Hubei
  - Local Institution - 007-701-Ph2, Changsha, Hunan
  - Hunan Cancer Hospital/Thoracic Medicine Department II, Changsha, Hunan
  - Local Institution - 1021-Ph2, Nanjing, Jiangsu
  - Local Institution - 1021, Nanjing, Jiangsu
  - Nanjing First Hospital/Department of Respiratory and Critical Care Medicine, Nanjing, Jiangsu
  - Nanjing First Hospital/Respiratory Department, Nanjing, Jiangsu
  - Local Institution - 1018-Ph2, Nanjing, Jiangsu
  - Local Institution - 1018, Nanjing, Jiangsu
  - Local Institution - 1020-Ph2, Nanjing, Jiangsu
  - Local Institution - 1020, Nanjing, Jiangsu
  - Local Institution - 1004-Ph2, Nantong, Jiangsu
  - Local Institution - 1004, Nantong, Jiangsu
  - Local Institution - 1017-Ph2, Xuzhou, Jiangsu
  - Local Institution - 1017, Xuzhou, Jiangsu
  - Local Institution - 007-713-Ph2, Nanchang, Jiangxi
  - Local Institution - 1040-Ph2, Nanchang, Jiangxi
  - Local Institution - 1040, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Local Institution - 1006-Ph2, Changchun, Jilin
  - Local Institution - 1006, Changchun, Jilin
  - Local Institution - 007-717-Ph2, Changchun, Jilin
  - The First Bethune Hospital Of Jilin University/Oncology Department, Changchun, Jilin
  - Local Institution - 007-741-Ph2, Shenyang, Liaoning
  - Local Institution - 007-741, Shenyang, Liaoning
  - Local Institution - 1008-Ph2, Shenyang, Liaoning
  - Local Institution - 1008, Shenyang, Liaoning
  - Local Institution - 007-749, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Local Institution - 007-702-Ph2, Shenyang, Liaoning
  - Local Institution - 007-702, Shenyang, Liaoning
  - Local Institution - 007-746-Ph3, Yinchuan, Ningxia
  - Local Institution - 007-746, Yinchuan, Ningxia
  - Local Institution - 007-718-Ph2, Xi'an, Shaanxi
  - Local Institution - 007-721-Ph2, Xi'an, Shaanxi
  - Local Institution - 007-721, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University/Medical Oncology Department, Xi'an, Shaanxi
  - Local Institution - 007-708-Ph2, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - Local Institution - 007-737-Ph2, Linyi, Shandong
  - Linyi Cancer Hospital/Oncology Department, Linyi, Shandong
  - Local Institution - 007-703-Ph2, Linyi, Shandong
  - Local Institution - 007-703, Linyi, Shandong
  - Local Institution - 007-709-Ph2, Shanghai, Shanghai Municipality
  - Local Institution - 007-709, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital-Oncology department, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center/Thoracic Oncology Department, Shanghai, Shanghai Municipality
  - Local Institution - 007-024-Ph2, Shanghai, Shanghai Municipality
  - Local Institution - 007-024-Ph3, Shanghai, Shanghai Municipality
  - Local Institution - 007-024, Shanghai, Shanghai Municipality
  - Local Institution - 007-035-Ph2, Shanghai, Shanghai Municipality
  - Local Institution - 007-740-Ph2, Taiyuan, Shanxi
  - Local Institution - 007-740, Taiyuan, Shanxi
  - Local Institution - 007-748, Taiyuan, Shanxi
  - Shanxi Provincial Cancer Hospital/Respiratory Medicine, Taiyuan, Shanxi
  - Local Institution - 007-710-Ph2, Chengdu, Sichuan
  - Local Institution - 007-710, Chengdu, Sichuan
  - Local Institution - 007-720-Ph2, Chengdu, Sichuan
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Local Institution - 007-711-Ph2, Luzhou, Sichuan
  - Local Institution - 007-711, Luzhou, Sichuan
  - Xinjiang Medical University Cancer Hospital - Urumqi, Ürümqi, Xinjiang
  - Local Institution - 007-743, Ürümqi, Xinjiang
  - Local Institution - 1036-Ph2, Ürümqi, Xinjiang
  - Local Institution - 1036, Ürümqi, Xinjiang
  - Local Institution - 1032-Ph2, Kunming, Yunnan
  - Local Institution - 1032, Kunming, Yunnan
  - Local Institution - 007-385-Ph3, Kunming, Yunnan
  - Local Institution - 007-385, Kunming, Yunnan
  - Local Institution - 007-745-Ph2, Kunming, Yunnan
  - Local Institution - 007-745, Kunming, Yunnan
  - Local Institution - 007-716-Ph2, Hangzhou, Zhejiang
  - Local Institution - 007-716, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Local Institution - 007-036-Ph2, Hangzhou, Zhejiang
  - Local Institution - 007-036, Hangzhou, Zhejiang
  - Local Institution - 007-037-Ph2, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Local Institution - 1050-Ph2, Taizhou, Zhejiang
  - Local Institution - 1050, Taizhou, Zhejiang
  - Taizhou Hospital Of Zhejiang Province, Taizhou, Zhejiang
  - Local Institution - 1043-Ph2, Qingdao
  - Local Institution - 1043, Qingdao
  - Local Institution - 007-035, Shanghai
- Colombia (2):
  - Local Institution - Unk021, Medellín
  - Local Institution - Unk027, Montería
- Croatia (3):
  - Local Institution - 007-4000, Pula
  - Specijalna Bolnica Medico, Rijeka
  - Local Institution - 007-4002, Zagreb
- Czechia (5):
  - Multiscan - Ambulance klinicke onkologie se stacionarem - Horovice, Hořovice
  - Fakultni Nemocnice Olomouc, Olomouc
  - Nemocnice AGEL Ostrava-Vitkovice, Ostrava
  - Local Institution - 007-163, Prague
  - Fakultni nemocnice Bulovka, Praha 8 - Liben
- Denmark (3):
  - Local Institution - 007-172, Odense
  - Sjukhus Sonderjylland, Sønderborg
  - Sygehus Lillebaelt - Vejle Sygehus, Vejle
- Finland (2):
  - Docrates Cancer Center, Helsinki
  - Tampereen Yliopistollinen Sairaala (TAYS), Tampere
- France (19):
  - Institut de Cancerologie de lOuest - Angers, Angers
  - Hopital Ambroise-Pare, Boulogne-Billancourt
  - Hopital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Hopital Michallon, La Tronche
  - Centre Hospitalier Universitaire Limoges, Limoges
  - Local Institution - 007-1993, Lorient
  - Local Institution - 007-199, Marseille
  - Hopital Nord de Marseille, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Hopital Emile Muller, Mulhouse
  - Local Institution - 007-664, Paris
  - Local Institution - 007-1991, Rennes
  - Centre Hospitalier Universitaire De Nantes - Hopital Nord Laennec, Saint-Herblain
  - Institut de Cancerologie de lOuest - Saint-Herblain - Site Rene Gauducheau, Saint-Herblain
  - Les Hopitaux Universitaires de Strasbourg, Strasbourg
  - Hopital Bretonneau, Tours
  - Local Institution - 007-202, Villejuif
- Georgia (6):
  - Local Institution - 007-790, Batumi
  - Local Institution - 007-065, Tbilisi
  - Local Institution - 007-795, Tbilisi
  - Local Institution - 007-789, Tbilisi
  - Local Institution - 007-063, Tbilisi
  - Institute of Clinical Oncology - Tbilisi, Tbilisi
- Germany (32):
  - Local Institution - 007-211A, Immenstadt im Allgäu, Bavaria
  - Local Institution - 007-675, Amberg
  - Local Institution - 007-2222, Augsburg
  - Local Institution - Link, M., Bad Homburg
  - Local Institution - Eggers, H., Braunschweig
  - Klinikum Chemnitz, Chemnitz
  - Local Institution - 007-2217, Cologne
  - Klinikum Esslingen, Esslingen am Neckar
  - Krankenhaus Nordwest, Frankfurt am Main
  - Universitatsklinikum Gieen und Marburg - Gieen, Giessen
  - LungenClinic Grosshansdorf, Grohansdorf
  - Asklepios Kliniken Barmbek, Hamburg
  - Local Institution - 007-2229, Hanover
  - Local Institution - 007-677, Heidelberg
  - Local Institution - 007-673, Heilbronn
  - Lungenklinik Hemer, Hemer
  - Local Institution - 007-225, Jena
  - Local Institution - 007-2225, Kaiserslautern
  - Klinikum Kassel, Kassel
  - Klinikverbund Allgau - Klinikum Kempten, Kempten
  - SLK-Kliniken - Fachklinik Lowenstein, Löwenstein
  - Universitatsklinikum Schleswig-Holstein - Campus Lubeck, Lübeck
  - Local Institution - 007-223, Mainz
  - Local Institution - 007-2221, Mönchengladbach
  - Local Institution - 007-2228, München
  - Munchen Klinik Bogenhausen, München
  - Local Institution - 007-2218, Neuruppin
  - Sana Klinikum Offenbach, Offenbach
  - Pius-Hospital Oldenburg, Oldenburg
  - Local Institution - 007-2226, Treuenbrietzen
  - Local Institution - 007-2227, Trier
  - Bundeswehrkrankenhaus Ulm, Ulm
- Greece (9):
  - Henry Dunant Hospital Center, Athens, Attica
  - General Hospital for Thoracic Diseases Sotiria, Athens
  - "General Hospital of Athens "Alexandra"", Athens
  - "University General Hospital "Attikon" - General Hospital of West Attica "H Agia Varvara"", Athens
  - University General Hospital of Heraklion (PAGNI), Heraklion
  - University General Hospital of Larissa, Larissa
  - "General Oncology Hospital of Kifisias "Agioi Anargyroi"", Nea Kifissia
  - Metropolitan Hospital, Piraeus
  - Saint Lukes Hospital, Thessaloniki
- Hong Kong (4):
  - Humanity & Health Clinical Trial Centre, Central
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Queen Mary Hospital - Hong Kong, Hong Kong
  - Queen Elizabeth Hospital - Hong Kong, Kowloon
- Hungary (7):
  - Semmelweis Egyetem - Pulmonologiai Klinika, Budapest
  - Orszagos Koranyi Pulmonologiai Intezet, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű
  - Matrai Gyogyintezet, Gyöngyös
  - Local Institution - 007-057, Tatabánya
  - Reformatus Pulmonologiai Centrum, Törökbálint
- India (22):
  - CIMS Hospital, Ahemdabad
  - Local Institution - 007-1574, Ahmedabad
  - Marathwada Cancer Hospital & Research Institute, Aurangabad
  - Local Institution - 007-1586, Bangalore
  - Local Institution - 007-1575, Belagavi
  - Local Institution - 007-1587, Howrah
  - Local Institution - 007-1564, Hyderabad
  - Basavatarakam Indo American Cancer Hospital & Research Institute, Hyderabad
  - Local Institution - 007-1569, Jaipur
  - Local Institution - 007-1566, Kochi
  - Netaji Subhas Chandra Bose Cancer Hospital & Research Institute, Kolkata
  - Meenakshi Mission Hospital and Research Centre, Madurai
  - Local Institution - Shetty, R., Mangalore
  - Tata Memorial Centre - Tata Memorial Hospital, Mumbai
  - Mysore Medical College and Research Institute, Mysore
  - Local Institution - 007-1588, New Delhi
  - Indraprastha Apollo Hospitals, New Delhi
  - Local Institution - 007-1578, New Delhi
  - Indira Gandhi Institute of Medical Sciences, Patna
  - Local Institution - 007-1571, Pune
  - Nirmal Hospital Pvt. Ltd., Rajkot
  - Local Institution - 007-1581, Varanasi
- Ireland (7):
  - Local Institution - 007-256, Cork
  - Beaumont Hospital - Dublin, Dublin
  - St. Jamess Hospital, Dublin
  - Tallaght University Hospital, Dublin
  - University Hospital Galway, Galway
  - Local Institution - 007-258, Limerick
  - University Hospital Waterford, Waterford
- Israel (9):
  - Emek Medical Center, Afula
  - Rambam Health Care Campus, Bat Galim
  - Soroka Medical Center, Beersheba
  - Local Institution - 007-263, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Ziv Medical Center, Zsfat
- Italy (23):
  - Local Institution - Unk016, Aviano
  - Istituto Tumori Bari Giovanni Paolo II - IRCCS, Bari
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico Sant Orsola-Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia, Brescia
  - Istituto di Candiolo - Fondazione del Piemonte per lOncologia, Candiolo
  - Azienda Ospedaliero - Universitaria Careggi, Florence
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale Policlinico San Martino, Genova
  - "Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST", Meldola
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) - Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan
  - Local Institution - 007-318, Monza
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Local Institution - Unk017, Padua
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Azienda Ospedaliera di Perugia - Santa Maria della Misericordia, Perugia
  - Azienda Sanitaria Territoriale Pesaro Urbino, Pesaro
  - Ospedale Santa Maria delle Croci di Ravenna, Ravenna
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Local Institution - Unk030, Rozzano
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Japan (17):
  - National Hospital Organization - Nagoya Medical Center, Nagoya, Aichi-ken
  - Jcho Chukyo Hospital, Nagoya, Chiba
  - Ehime University Hospital, Toon-shi, Ehime
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Local Institution - 007-1593, Nishinomiya-Shi, Hyōgo
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Nara Medical University Hospital, Kashihara, Nara
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai-Shi, Osaka
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni
  - Kanazawa University Hospital, Kanazawa
  - Kochi Medical School Hospital, Nankoku-shi
  - Osaka City General Hospital, Osaka
  - Osaka Prefectural Hospital Organization - Osaka International Cancer Institute, Osaka
  - Local Institution - 007-1164, Toyama
- Malaysia (8):
  - Local Institution - Unk079, Johor Bahru, Johor
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Local Institution - Choo Khoon, O., George Town, Pulau Pinang
  - Local Institution - Unk048, George Town, Pulau Pinang
  - Local Institution - Unk007, Petaling Jaya, Selangor
  - Sunway Medical Centre, Petaling Jaya, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Local Institution - Unk075, Kuala Lumpur
- Mexico (8):
  - Local Institution - 007-476, Guadalajara, Jalisco
  - Local Institution - Unk070, Guadalajara, Jalisco
  - Local Institution - Unk034, Mexico City, Mexico City
  - Local Institution - Unk049, Mexico City, Mexico City
  - Local Institution - 007-475, Mexico City
  - Local Institution - Unk037, Monterrey
  - Local Institution - 007-477, Monterrey
  - Local Institution - Unk026, Monterrey
- Netherlands (9):
  - Het Nederlands Kanker Instituut, Amsterdam
  - Albert Schweitzer Ziekenhuis - Dordwijk, Dordrecht
  - Local Institution - 007-303, Harderwijk
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Franciscus Gasthuis & Vlietland - Gasthuis, Rotterdam
  - Local Institution - 007-308, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Local Institution - 007-305, Zwolle
- Health New Zealand - Te Whatu Ora - MidCentral, Palmerston North, New Zealand
- Local Institution - 007-310, Drammen, Norway
- Peru (12):
  - Local Institution - Unk080, Trujillo, La Libertad
  - Local Institution - Unk022, Jesus Maria, Lima region
  - Local Institution - Unk031, Lima Cercado, Lima region
  - Local Institution - Unk024, Miraflores, Lima region
  - Local Institution - Unk042, San Isidro, Lima region
  - Local Institution - Unk071, San Isidro, Lima region
  - Local Institution - Unk054, Surquillo, Lima region
  - Local Institution - Unk051, Arequipa
  - Local Institution - Unk023, Arequipa
  - Local Institution - Unk044, Arequipa
  - Local Institution - Unk040, Cusco
  - Local Institution - Unk046, Lima
- Philippines (6):
  - Local Institution - 007-1541, Bacolod City
  - Local Institution - 007-1545, Cebu City
  - Local Institution - 007-1544, Iloilo City
  - Local Institution - 007-1543, Makati City
  - Local Institution - 007-1542, Molo
  - Local Institution - 007-1540, Quezon City
- Poland (11):
  - Uniwersyteckie Centrum Kliniczne w Gdansku, Gdansk
  - Swietokrzyskie Centrum Onkologii Samodzielny Publiczny Zaklad Opieki Zdrowotnej w Kielcach, Kielce
  - Pratia MCM Krakow, Krakow
  - MS Pneumed - Janusz Milanowski, Katarzyna Szmygin-Milanowska Spolka Jawna, Lublin
  - Warminsko-mazurskie Centrum Chorob Pluc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc I Gruzlicy, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii im. Eugenii i Janusza Zeylandow, Poznan
  - Pratia Poznan, Skorzewo
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
  - Local Institution - 007-056, Warsaw
  - Local Institution - 007-322, Warsaw
- Portugal (9):
  - Unidade Local de Saude de Coimbra, Coimbra
  - Unidade Local de Saude do Alto Ave, E. P. E (Hospital da Senhora da Oliveira Guimaraes), Guimarães
  - Instituto Portugues De Oncologia De Lisboa Francisco Gentil, Lisbon
  - Local Institution - 007-338-A, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Hospital CUF Porto, Porto
  - Unidade Local de Saude de Santo Antonio, E. P. E - Hospital Geral de Santo Antonio, Porto
  - Local Institution - 007-339, Porto
  - Local Institution - 007-335, Vila Nova de Gaia
- Romania (5):
  - Institutul Oncologic Bucuresti - Prof. Dr. Alexandru Trestioreanu, Bucharest
  - Medisprof, Cluj-Napoca
  - Centrul de Radioterapie Amethyst Cluj, Floreşti
  - Centrul de Oncologie Euroclinic, Iași
  - Oncocenter - Oncologie Clinica, Timișoara
- Serbia (4):
  - Univerzitetski Klinicki Centar Srbije, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - Local Institution - 007-694, Kragujevac
  - Uzice General Hospital, Užice
- Singapore (2):
  - Raffles Hospital, Singapore
  - Curie Oncology - Farrer - 10-05, Singapore
- South Africa (3):
  - Local Institution - 007-4010, Port Elizabeth, Eastern Cape
  - Local Institution - 007-4013, Johannesburg, Gauteng
  - Local Institution - 007-4012, Pretoria, Gauteng
- South Korea (12):
  - Inje University Haeundae Paik Hospital, Busan
  - Pusan National University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center - Korea, Goyang-si
  - Inha University Hospital, Junggu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Catholic University of Korea St. Vincents Hospital, Suwon
- Spain (24):
  - Local Institution - 007-611 A, Pamplona, Navarre
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Institut Catala dOncologia Badalona, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall dHebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Local Institution - Unk081, Bilbao
  - Local Institution - Unk063, Burgos
  - Local Institution - Unk014, Jerez de la Frontera
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria
  - Local Institution - Unk012, León
  - Institut Catala dOncologia - Hospital Duran i Reynals (ICO LHospitalet), LHospitalet de Llobregat
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga - Hospital Civil, Málaga
  - Local Institution - 007-604, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Local Institution - Unk013, Gävle, Sweden
- Switzerland (2):
  - Local Institution - 007-397, Sankt Gallen
  - Local Institution - 007-396, Villars-sur-Glâne
- Taiwan (9):
  - Local Institution - 007-127, Taichung
  - Local Institution - 007-128, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital - Liouying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Taipei Medical University - Shuang Ho Hospital, Ministry of Health and Welfare, Taipei
  - Chang Gung Memorial Hospital - Linkou Branch, Taoyuan District
- Thailand (2):
  - Local Institution - 007-139, Bangkok
  - Local Institution - Runglodvatana, Y., Bangkok
- Turkey (Türkiye) (21):
  - Baskent Universitesi Adana Uygulama Ve Arastirma Hastanesi, Alanya
  - T.C. Saglik Bakanligi - Istanbul Il Saglik Mudurlugu - Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Altındağ
  - Hacettepe Universitesi Kanser Enstitusu, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Liv Hospital Ankara, Ankara
  - Local Institution - 007-3810, Antalya
  - VM Medical Park Samsun Hastanesi, Atakum
  - Memorial Bahcelievler Hospital, Bahçelievler
  - Ege Universitesi Tip Fakultesi Hastanesi, Bornova
  - T.C. Saglik Bakanligi Ankara Bilkent Sehi�r Hastanesi�, Çankaya
  - Trakya Universitesi Tip Fakultesi, Edirne
  - Istanbul Universitesi Onkoloji Enstitusu, Fatih
  - Ozel Gaziantep Medical Point Hastanesi, Gaziantep
  - Local Institution - 007-069, Istanbul
  - Istanbul Onkoloji Hastanesi, Istanbul
  - Izmir Ekonomi Universitesi Medical Point Hastanesi, Izmir
  - Yeditepe Universitesi Kosuyolu Hastanesi, Kadıköy
  - Kocaeli Universitesi Arastirma ve Uygulama Hastanesi, Kocaeli
  - Inonu Universitesi Turgut Ozal Tip Merkezi, Malatya
  - Ankara Universitesi Tip Fakultesi - Cebeci Arastirma ve Uygulama Hastanesi, Mamak
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Hastanesi, Şişli
- United Kingdom (8):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Local Institution - 007-415, Edinburgh
  - Local Institution - 007-403, Kent
  - University Hospitals of Leicester NHS Trust, Leicester
  - University College London Hospitals NHS Foundation Trust, London
  - Guys and St Thomas NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Surrey County Hospital NHS Foundation Trust, Surrey

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04613596.html